CLINICAL TRIAL: NCT03998774
Title: Uncontrolled Prospective Monocentric Study Aiming to Evaluate the Anxiolytic Effect of EMONO in Children During Dental Care
Brief Title: Evaluation Ofe the Anxiolytic Effect of EMONO in Children During Dental Care (MOPEA)
Acronym: MOPEA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0275
Record Dates: First submitted 2019-05-28; First posted 2019-06-26 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Dental Care for Children
Keywords: Nitrous oxide; Conscious sedation; Paediatric dentistry
MeSH Terms: interventions — Meopa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Evaluate the anxiolytic effect during dental care with MEOPA in children — Primary Purpose: The main objective of this study is to evaluate the anxiolytic effect of EMONO in children during dental care.
  Enrollment: 30

SUMMARY:
The EquiMolar Oxygen and Nitrous Oxyde mix (EMONO) is listed by the ANSM (National Agency for the Safety of Medicines and Health Products) as drugs with enhanced surveillance. EMONO is a gas composed equally of oxygen and nitrous oxide, presented in bottle. The University Hospital of Nantes is currently conducting a general evaluation of the EMONO use in the hospital context. The department of odontology is part of this movement and wants to study the anxiolytic effect expected during dental care under MEOPA in children in the Dental Care Center. This analysis follows a previous study (MEOPAeDent) that subjectively took into account this anxiolysis.

DETAILED DESCRIPTION:
The EquiMolar Oxygen and Nitrous Oxide Mix (EMONO) is listed by the ANSM (National Agency for the Safety of Medicines and Health Products) as drugs with enhanced surveillance. EMONO is a gas composed equally of oxygen and nitrous oxide, presented in bottle. It has had a marketing authorization in France since 2001. Until 2009, it was reserved for hospital use and emergency vehicles; and indicated in the analgesia of short-term painful acts or during medical assistance. urgency in adults and children, dental sedation in children and frail subjects, and obstetrics. The actual benefit was considered important by the Transparency Committee.

Since 2009, a modification of the MAH for EMONO-based specialties has authorized their release from the hospital reserve, which can now be issued for professional use in city and dental surgery. Given the risks associated with the use of EMONO, in particular its potential for abuse and dependence, the ANSM conditioned its availability outside health facilities to the implementation of a common national RMP. This measure was also accompanied by a national monitoring of pharmacovigilance and addictovigilance. The latter is under the responsibility of CEIP-A of Nantes.

The University Hospital of Nantes is currently conducting a general evaluation of the use of EMONO in the hospital context. The department of odontology is part of this movement and wants to study the anxiolytic effect expected during dental care under EMONO in children in the Dental Care Center. This analysis follows a previous study (MEOPAeDent) that subjectively took into account this anxiolysis.

The analysis of this study will allow us to improve the good use of MEOPA for dental care.

ELIGIBILITY:
Inclusion Criteria:

* Children from 3 to 15 years,
* Requiring dental treatment under EMONO including local anesthesia
* Not opposed, as well as parents, to participate in the study
* Having a sufficiently cooperative attitude to allow the installation of the monitoring equipment
* The use of EMONO for dental care must be a first time for the child

Exclusion Criteria:

* The excluded patients will be those whose number of care is too important, justifying a general anesthesia. Similarly, patients who do not require anesthesia for their care will be excluded.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from 3 to 15 years old, requiring MEOPA treatment with local anaesthesia for the first time
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the anxiolytic effect of EMONO in children during dental care | 15 minutes
  The primary endpoint will be a significant variation of heart rate at 3 key moments of the treatment session:
  * Chair installation
  * 5 minutes after induction of MEOPA induction
  * The injection of the local anesthetic

SECONDARY OUTCOMES:
Assess whether the child's stress is less intense after certain types of dental care under EMONO by the measure of heart rate variation. | 1 minute
  The criterion for assessing the child's stress based on the care taken will be the significant variation in heart rate at another point in the treatment session: at the time of the end of the inhalation and care. Comparison will be made between children having pulptomy or extraction.
Assess whether the child's stress is less intense after certain types of dental care under EMONO by the measure Veerkamp Modified VENHAM Anxiety Assessment Scale. | 1 minute
  A Veerkamp Modified VENHAM Anxiety Assessment Scale will also be used before and after dental care ( from 0 to relaxed to 5 for extremely stressed) by the dentist. Comparison will also be made between chidren having pulpotomy or extraction.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Prud'homme, Principal Investigator — Nantes University Hospital
Locations (1):
- Chu de Nantes, Nantes, France